CLINICAL TRIAL: NCT04533308
Title: The Impact of Virtual Reality on the Emotional State of Patients With Aphasia During Rehabilitation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Eduard Novak, MD, MSc, State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMSC-02-20
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Aphasia; Virtual Reality; Emotional Disturbances
MeSH Terms: conditions — Aphasia; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR intervention (Experimental): Participants will have a session in VR for 20-30 minutes each working day. They can choose natural 360-degrees scenes from different locations in the world with or without interactions with animals. The equipment will include HTC Vive (HTC Corporation).
  Interventions: Behavioral: Relaxation in virtual reality
- Control (No Intervention): Patients in the control group will not receive any psychological interventions.

INTERVENTIONS:
Behavioral: Relaxation in virtual reality — Natural 360-degrees scenes from different locations in the world with or without interactions with animals in the virtual reality
  Arms: VR intervention

SUMMARY:
The aim of the study is to determine virtual reality (VR) impact during standard program of rehabilitation on emotional state of patients with aphasia.

DETAILED DESCRIPTION:
Aim 1: To test the safety of virtual reality in a vulnerable population of patients with aphasia during rehabilitation. Participants will be alternately assigned to receiving a relaxation session in VR every working day during a standard course of rehabilitation.

Aim 2: To test the preliminary efficacy of combining VR with the course of rehabilitation to promote emotional improvements in patients with aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate aphasia of any type
* Russian is primary language
* At least 2 weeks post cardio-vascular accident (ischemic or hemorrhagic stroke) or head injury of any location
* Have a history of only one stroke
* Medically stable

Exclusion Criteria:

* Associated severe cognitive deficits and psychiatric disorders which prevent patients understanding of the informed consent
* Epilepsy
* Medical history of severe visual or hearing impairment
* Comorbid neurological diagnosis (e.g. epilepsy, multiple sclerosis, Parkinson disease, dementia)
* Unable to perform the required exercises due to severe motor, sensory or cognitive deficit (memory, attention, executive functioning, apraxia, regulatory and planning activities etc.) and medical problems (for example, anyone meeting New York Heart Association Class IV criteria, hospitalization for myocardial infarction or heart surgery within 120 days, severe cardiomyopathy or documented serious and unstable cardiac arrhythmias)
* Drug or alcohol addiction within the last 6 months.
* Significant current psychiatric illness defined as affective disorder unresponsive to medication or bipolar affective disorder, psychosis, schizophrenia or suicidality
* Current participation in another interventional trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The absence of severe adverse reactions | From admission to discharge, up to 3 weeks
  Assessed by a self-reported form and physiological parameters

SECONDARY OUTCOMES:
10 - Stroke Aphasic Depression Questionnaire (SADQH-10) | From admission to discharge, up to 3 weeks
  Scores range from 0 to 30 with lower scores denoting better outcomes.
Visual Analog Mood Scale (VAMS) | From admission to discharge, up to 3 weeks
  Scores range from 0 to 10 with lower scores denoting better outcomes.
Perceived Stress Scale (PSS) | From admission to discharge, up to 3 weeks
  Scores range from 0 to 50 with lower scores denoting better outcomes.
Three-level European quality of life five-dimensional questionnaire | From admission to discharge, up to 3 weeks
  There are five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Patients choice results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describe the health status.
Aphasic Depression Rating Scale (ADRS) | From admission to discharge, up to 3 weeks
  Scores range from 0 to 36 with lower scores denoting better outcomes.
Lüscher Color Test | From admission to discharge, up to 3 weeks
  Eight different colored cards are place in order of preference. The descriptive statements formed by Lüscher for each color were used to interpret the results.

CONTACTS AND LOCATIONS:
Overall Officials: Vadim D Daminov, Prof, Principal Investigator — Pirogov National Medical and Surgical Center
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 1 year after completion of the trial
Access Criteria: upon request